CLINICAL TRIAL: NCT00500591
Title: Prevalence of Endometrial Abnormalities In Obese Women
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0018
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Obesity
Keywords: Endometrial Abnormalities; Endometrial Cancer; Obesity; Survey; Questionnaire
MeSH Terms: conditions — Obesity; Endometrial Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples used to look at different hormone levels related to risk of endometrial abnormalities. An endometrial biopsy will be performed to collect a tissue sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese Women
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire regarding weight history, gynecologic, and medical history, lasting about 30 minutes.
  Other Names: Survey

SUMMARY:
It is known that women who are obese are at higher risk of endometrial cancer (cancer of the lining of the uterus or womb). The goal of this clinical research study is to find out how common abnormalities of the endometrium are in women who are considered obese and to find out if those same abnormalities are less common in women who are considered to be thin. Researchers would like to learn if obese patients have symptoms (like irregular menstrual cycles) that may mean there could be an abnormality present. Researchers would also like to know if obese women have access to regular female exams and whether they routinely go to their primary care doctors.

DETAILED DESCRIPTION:
Women in this study will be asked to complete three different parts of the study. All three parts of the study will be done during one visit to the gynecology center. First, you will be asked to complete a survey/questionnaire that will give researchers information on your background, weight history, gynecologic, and medical history. You will be assisted by a research nurse and completion of the questionnaire is expected take about 30 minutes.

Second, you will be asked to have a blood sample drawn. About 2 tablespoons of blood will be drawn. This blood will be used to look at different hormone levels that may be related to your risk of endometrial abnormalities.

Third, an endometrial biopsy will be performed by one of the doctors running the study. This will require you to have a full pelvic exam (much like when you have a pap smear), which will include looking at the cervix (mouth of the womb) and putting a small pipelle (straw) into the womb to collect a tissue sample. This procedure is routinely done in the office. You will not be required to take medications prior to the procedure and you will not receive a prescription for pain medication once the procedure is complete.

Completion of all three parts of the study may take between one to two hours. You and your physician will be notified of your endometrial biopsy results.

This is an investigational study. Up to 200 participants will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a measured BMI greater than or equal to 30 kg/m2 (obese) or less than or equal to 25 kg/m2 (lean) at the time of enrollment.
2. Patients must be between the ages of 30 and 55 years old at the time of enrollment.
3. Patients must not have taken any birth control (including pills, patch, injectables) for at least three months prior to enrollment.
4. Patients may not be pregnant at the time of enrollment (defined by negative urine pregnancy test).
5. Patients must have signed an informed consent indicating they are aware of the investigational nature of this study.
6. Patients with a history of non-metastatic cancer may be included if they have not undergone cancer treatment for at least six months prior to enrollment.

Exclusion Criteria:

1. Patients who have had a prior hysterectomy.
2. Patients who are pregnant or have a positive pregnancy test.
3. Patients with a prior history of endometrial hyperplasia or endometrial cancer.
4. Patients who are currently on birth control (including pills, patch, or injectable birth control).
5. Patients who are postmenopausal (have not had a menstrual cycle in greater than or equal to one year).
6. Patients who have ever been on selective estrogen receptor modulators (SERMs) in the past including Tamoxifen and Raloxifene.
7. Patients with a history of metastatic cancer (any type).
8. Patients with a history of non-metastatic cancer who are currently undergoing therapy for that cancer or who have received therapy within six months of enrollment.
9. Patients with a history of non-metastatic cancer who have received any type of hormonal therapy including but not limited to aromatase inhibitors, GNRH-agonists, and Zoladex.
10. Patients who have had prior radiation to the pelvis.
11. Patients with psychiatric disorders that would interfere with consent.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study participants with a measured BMI greater than or equal to 30 kg/m^2 (obese) or less than or equal to 25 kg/m^2 (lean) at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2004-06 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Endometrial Abnormalities in Obese and Lean Women | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Karen H. Lu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Dottino JA, Zhang Q, Loose DS, Fellman B, Melendez BD, Borthwick MS, McKenzie LJ, Yuan Y, Yang RK, Broaddus RR, Lu KH, Soliman PT, Yates MS. Endometrial biomarkers in premenopausal women with obesity: an at-risk cohort. Am J Obstet Gynecol. 2021 Mar;224(3):278.e1-278.e14. doi: 10.1016/j.ajog.2020.08.053. Epub 2020 Aug 21. PMID 32835719
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org